CLINICAL TRIAL: NCT02279030
Title: Three Dimensional Neuro-cardiac Imaging Using 123I-metaiodobenzylguanidine Single Photon Emission Computed Tomography to Guide Premature Ventricular Contractions Ablations
Brief Title: Use of MIBG Scan Images in PVC Ablations
Acronym: PVC-MIBG
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Timm-Michael Dickfeld, CARDIAC ELECTROPHYSIOLOGY PHYSICIAN, University of Maryland, Baltimore
Other Study IDs: HP-00062156
Record Dates: First submitted 2014-10-20; First posted 2014-10-30 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Premature Ventricular Contractions
Keywords: ablation
MeSH Terms: conditions — Ventricular Premature Complexes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: MIBG nuclear scan — To have scan to help define pathways for PVC ablations.
  Other Names: PVC ablations

SUMMARY:
The purpose of this study is to assess if Single Photon Emission Computed Tomography (SPECT) demonstrating cardiac innervation can be integrated into current electrophysiology voltage mapping system and provide improved guidance for ablation of PVCs.

DETAILED DESCRIPTION:
Premature ventricular contractions (PVC) are the most common arrhythmia to be observed in the absence of structural heart disease, and 'frequent' PVCs are estimated to occur in 1-4% of the general population.1 Idiopathic PVCs are usually associated with a benign course from the standpoint of arrhythmic death, but often result in significant symptoms for the patient such as palpitations, dizziness, pre-syncope and rarely syncope. More recently, a new concept of PVC- mediated cardiomyopathy has emerged that is reversible with suppression of the PVCs.2 Both of those patient populations are currently targeted with PVC suppressive therapy which often involves as the first step using medical therapy such as a beta blocker, calcium channel blocker or an antiarrhythmic. If those fail or if the patients wants to avoid medical therapy an ablation to eliminate the abnormal myocardial tissue that is the origin of the PVCs is often performed.

Radiofrequency ablation (RFA) for PVCs has been performed for several decades and has a well-defined safety and effectiveness profile in patients with symptomatic frequent ventricular ectopic beats and PVC-induced cardiomyopathy. Successful PVC suppression ≥80% of RV and LV PVCs has been reported to be as high as ~80% using an ablation approach.9 Studies found improvements in patient symptoms with elimination of PVCs. In LV dysfunction following ablation demonstrated a significant inverse correlation between EF and PVC burden before ablation, and a significant post procedural improvement in ejection fraction (EF) in 82% of patients who had abnormal systolic function before ablation.8 Improvement of the overall LV EF ranged from 13%-23% after PVC ablation.5,8,10

Autonomic innervation of the heart plays a major role in the normal regulation of myocardial function, heart rate, and coronary blood flow. Abnormal sympathetic cardiac innervation has been shown to have prognostic value for different heart diseases, e.g. heart transplant, coronary artery disease, heart failure, arrhythmias, etc. Importantly, there is a clear association with an increased cardiac morbidity and mortality in heart diseases. Patients with myocardial infarction as well as patients with heart failure exhibit well recognized abnormalities in autonomic tone. PVCs especially in the setting of preserved EF (normal heart patients) have frequently an automatic/triggered mechanism, which is influenced by the cardiac innervation.

Decreased reuptake by impaired myocardial presynaptic nerve terminals results in a buildup of these catecholamines in the synaptic cleft. This leads to a downregulation of postsynaptic beta-adrenergic receptors, with resultant worsening cardiomyopathy and increased arrhythmogenesis.

Cardiac sympathetic innervation can be directly imaged with commonly used nuclear radioisotope, 123I-meta-iodobenzylguanidine (123I-mIBG). As a norepinephrine analogue, 123I-mIBG is similarly released into the synaptic cleft in response to sympathetic input by presynaptic nerve terminals 123I-metaiodobenzylguanidine (123I-MIBG) allows visualization of the cardiac innervation, which could provide additional information to understand the origin, prognosis and pathophysiology of PVCs and guide potential ablation procedures.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for PVC ablation

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients requiring PVC ablation
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-06; Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Utilization of MIBG imaging for PVC ablations | 2 years
  To determine if MIBG imaging provides decreased PVC ablation time
Decrease PVC occurrence | 2 years
  Does MIBG imaging allow for treatment that provides improved outcomes in decreasing PVCs
Increase in Motility | 2 years
  Do MIBG follow-ups demonstrate an improvement in cardiac motility

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States